CLINICAL TRIAL: NCT05844904
Title: Mapping of Indonesians' Skin Type Based on Baumann Skin Type Indicator-Indonesia (BSTI-Ina) Questionnaire and Development of Artificial Intelligence Modelling BSTI-Ina: A Multicentric Study
Brief Title: Mapping of Indonesians' Skin Type Based on Baumann Skin Type Indicator-Indonesia and Development of Artificial Intelligence Modelling
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Dr.dr.Irma Bernadette, SpKK (K) (Other)
Collaborators: Indonesian Society of Dermatology and Venereology (Unknown); College of Dermatologist and Venereologist (Unknown); Indonesia Medical Education and Research Institute (Other)
Responsible Party: Sponsor-Investigator, Dr.dr.Irma Bernadette, SpKK (K), Prof. Dr. dr. Irma Bernadette S. Sitohang, SpKK(K) - Head of Cosmetic Dermatology Division, Dermatology and Venereology Department, Faculty of Medicine, Universitas Indonesia, dr. Cipto Mangunkusumo Hospital, Jakarta, Indonesia, Indonesia University
Organization: Indonesia University (Other)
Other Study IDs: MappingofBSTI
Record Dates: First submitted 2023-04-05; First posted 2023-05-06 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Baumann Skin Type Indicator
Keywords: skin type; Baumann Skin Type Indicator; artificial intelligence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- General: This research is an observational study. There's no control and experimental group.

SUMMARY:
The goal of this observational study is to learn about the skin type of Indonesians based on Baumann Skin Type Indicator Questionnaire in Indonesian language version, and to develop artificial intelligence modelling of BSTI-Ina. The main questions it aims to answer are:

1. What is the measurement of the validity and reliability of BSTI-Ina questionnaire year 2006 version which was adapted from BSTI questionnaire in English language year 2006 version as a specific measurement to identify skin type?
2. What is the measurement of the validity and reliability of BSTI-Ina questionnaire year 2022 version which was adapted from BSTI questionnaire in English language year 2022 version as a specific measurement to identify skin type?
3. What is the comparison of the validity and reliability between BSTI-Ina questionnaire year 2006 and year 2022 to determine Indonesian adult population's skin type?
4. How is the mapping of Indonesians' skin type based on BSTI-Ina?
5. What is the proportion of each skin type based on BSTI-Ina in Indonesian population?
6. What is the proportion of each skin type based on BSTI-Ina in Indonesian population sociodemographically?
7. How can Artificial Intelligence help categorize skin type based on BSTI-Ina automatically?

Participants are males and females between 18-59 year old. Participants will be asked to fill BSTI-Ina questionnaire. Participants then will be photographed in five different positions.

DETAILED DESCRIPTION:
This research is an observational study with a cross-sectional design. The aims of this study is to determine the validity and reliability of BSTI questionnaire translated in Indonesian and to develop artificial intelligence modelling for BSTI-Ina based on photographs. This study will be held in 13 research centers with a total of 1950 subjects consists of males and females age 18-59. It conducts of 2 phases. Phase 1 is to determine which version of BSTI will be used based on which one is more valid and reliable being translated in Indonesian and will be conducted in Jakarta as a pilot. In phase 1, participants will be asked to fill both BSTI-Ina 2006 and 2002 questionnaire. Participants then will be photographed in five different positions. Data will be analyzed to determine which of BSTI-Ina version is more valid and reliable. After deciding which BSTI-Ina version will be used, the study then goes to phase 2. Phase 2 will be conducted in 12 other research centers in Indonesia to map Indonesian population skin type. In both 2 phases, all participants will be asked to fill in BSTI-Ina questionnaire (either 2006 or 2022 version based on the result of Phase 1). Participants then will be photographed in five different positions. After all the data from all research centers are collected, data will be analyzed to map Indonesian population's skin type. Data as participants' skin types and photographs will also be processed by machine to model artificial intelligence. The aim is to automatically categorize skin type based on BSTI-Ina based on photographs.

ELIGIBILITY:
Inclusion Criteria:

* Males and females age 18-59 year old.
* Fitzpatrick's skin type III-V
* Educational degree of minimum high school
* Can speak Indonesian
* Can read
* Willing to participate and sign informed consent

Exclusion Criteria:

* Participant who doesn't fill the questionnaire completely
* Participant with skin disease involving >25% facial area

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: General adult population
Sampling Method: Non-Probability Sample
Enrollment: 1950 (Estimated)
Dates: Start 2023-09-08 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Baumann Skin Type Indicator questionnaire 2006 version in Indonesian language | Up to 2 weeks
  Adapting Baumann Skin Type Indicator questionnaire 2006 version to Baumann Skin Type Indicator questionnaire 2006 version in Indonesian language by certified translators
Baumann Skin Type Indicator questionnaire 2022 version in Indonesian language | Up to 2 weeks
  Adapting Baumann Skin Type Indicator questionnaire 2022 version to Baumann Skin Type Indicator questionnaire 2022 version in Indonesian language by certified translators
More valid and reliable version of Baumann Skin Type Indicator-Ina questionnaire (2006 or 2022 version) | Up to 1 month
  Comparing between Baumann Skin Type Indicator-Ina questionnaire 2006 version and 2022 version by statistician
Mapping of Indonesian population's skin type based on Baumann Skin Type Indicator-Ina | Up to 2 months
  Determine the proportion of Indonesia population's skin type based on Baumann Skin Type Indicator in 13 research centers
Capability of artificial intelligence model to categorize skin type based on Baumann Skin Type Indicator-Ina | Up to 1 month
  Data such as participants' skin types and photographs will be analyzed by machine resulting AI to categorize skin type automatically by photographs.

CONTACTS AND LOCATIONS:
Overall Officials: Irma Bernadette, MD, Principal Investigator — Faculty of Medicine, University of Indonesia; Hanny Nilasari, MD, Study Director — Faculty of Medicine, University of Indonesia; Sandra Widaty, MD, Study Director — Faculty of Medicine, University of Indonesia; Nelva K Jusuf, MD, Study Director — Faculty of Medicine, University of North Sumatra; Puguh Riyanto, MD, Study Director — Faculty of Medicine, Diponegoro University; Asnawi Madjid, MD, Study Director — Faculty of Medicine, Hasanuddin University; Marlyn G Kapantow, MD, Study Director — Faculty of Medicine, Sam Ratulangi University; I Gusti Ayu A Praharsini, MD, Study Director — Faculty of Medicine, Udayana University; Reti Hindritiani, MD, Study Director — Faculty of Medicine, Padjadjaran University; Diah M Indramaya, MD, Study Director — Faculty of Medicine, Airlangga University; Yuli Kurniawati, MD, Study Director — Faculty of Medicine, Sriwijaya University; Satya W Yenny, MD, Study Director — Faculty of Medicine, Andalas University; Arie Kusumawardani, MD, Study Director — Faculty of Medicine, Sebelas Maret University; Shinta Murlistyarini, MD, Study Director — Faculty of Medicine, Brawijaya University; Flandiana Yogianti, MD, Study Director — Faculty of Medicine, Gadjah Mada University; Aria Kekalih, MD, Study Director — Faculty of Medicine, University of Indonesia; Prasandhya A Yusuf, PhD, Study Director — Indonesia Medical Education and Research Institute, University of Indonesia; Eric D Tenda, MD, Study Director — Indonesia Medical Education and Research Institute, University of Indonesia; Vanya V Valindria, PhD, Study Director — Indonesia Medical Education and Research Institute, University of Indonesia; Sari Chairunnisa, MD, Study Director — Paragon Technology & Innovation; Irwan Batubara, MD, Study Director — Faculty of Medicine, University of Indonesia
Locations (13):
- Indonesia (13):
  - Rumah Sakit Umum Pusat Prof. Dr. I Goesti Ngoerah Gde Ngoerah, Denpasar, Bali
  - Rumah Sakit Umum Pusat Dr. Kariadi, Semarang, Central Java
  - Rumah Sakit Umum Daerah Dr. Moewardi, Surakarta, Central Java
  - Rumah Sakit Umum Pusat Nasional Dr. Cipto Mangunkusumo, Jakarta Pusat, DKI Jakarta
  - Rumah Sakit Umum Daerah Dr. Saiful Anwar, Malang, East Java
  - Rumah Sakit Umum Daerah Dr. Soetomo, Surabaya, East Java
  - Rumah Sakit Umum Pusat Prof. dr. R. D. Kandou, Manado, North Sulawesi
  - Rumah Sakit Universitas Sumatera Utara, Medan, North Sumatra
  - Rumah Sakit Umum Pusat Dr. dr. Wahidin Sudirohusodo, Makassar, South Sulawesi
  - Rumah Sakit Umum Pusat Dr. Mohammad Hoesin, Palembang, South Sumatra
  - Rumah Sakit Umum Pusat Dr. Sardjito, Yogyakarta, Special Region of Yogyakarta
  - Rumah Sakit Umum Pusat Dr. Hasan Sadikin, Bandung, West Java
  - Rumah Sakit Umum Pusat Dr. M. Djamil, Padang, West Sumatra

IPD SHARING:
Plan to Share IPD: Undecided